CLINICAL TRIAL: NCT01835964
Title: Biobehavioral Mechanisms of Glucose Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Marc Breton, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16723
Record Dates: First submitted 2013-04-11; First posted 2013-04-19 (Estimated); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Glucose Variability (GV); Continuous Glucose Monitor (CGM); Average Daily Risk Range (ADRR); Self Monitoring Blood Glucose (SMBG)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glucose Variability Observation (Experimental): The study procedures will start after CGM device training & practice using the blinded CGM for 2 days and will continue over the course of ~33 days. The study team will collect data about diabetes management including blood glucose data from fingerstick and CGM values along with insulin pump records throughout the 4 week observation period. Insulin sensitivity will be evaluated at home with predetermined meals' carbohydrate count. At the mid-study point glucose variability will be simulated in clinic with a metabolic challenge (liquid mixed meal) followed 4 hours later by the induction of hypoglycemia with an intravenous insulin injection. Insulin sensitivity, as well as glucagon and epinephrine counterregulatory responses will be evaluated to be related to overall Glucose Variability.
  Interventions: Procedure: Glucose Variability Observation

INTERVENTIONS:
Procedure: Glucose Variability Observation — On the morning of ~Day 17 for a metabolic challenge involving a standardized liquid mixed meal intended to raise the blood glucose approximately 150 mg/dl, followed four hours later by the induction of hypoglycemia with intravenous insulin administration with goal glucose of 55 mg/dl. After carbohydrate rescue, the subject will receive a meal and will be monitored until glucose is stable above 80 mg/dl.

SUMMARY:
The purpose of this study is to investigate how blood sugar changes in response to insulin and what the body does to counter-act low blood sugar in people with Type 1 Diabetes Mellitus. Insulin sensitivity is the term used to describe blood sugar changes within the body in response to insulin. Greater understanding of insulin sensitivity, particularly how the body responds to low blood sugar, will help us to better predict how blood sugar levels will change.

All subjects will receive a liquid mixed-meal and will have their blood sugar response monitored in order to study insulin sensitivity. All subjects will receive additional insulin injections that are given to cause a low blood sugar in order to understand how the body responds to a low blood sugar. All subjects will be closely monitored during the time the insulin is given, by frequent checks of blood sugar and constant medical and nursing supervision. Details of the visits, tests and procedures are described below. During this study, the study team will ask that subjects to use their own insulin pump and own glucometer. Subjects will need to use the same glucometer for the entire study. Subjects will be provided 1 box of strips. Subjects will be required to use lispro (Humalog) insulin 2-3 days before your inpatient admission which will be provided free of charge.

DETAILED DESCRIPTION:
Glucose variability (GV) in type 1 diabetes (T1DM) is increasingly viewed as a primary marker of glycemic control, responsible, along with chronic hyperglycemia reflected by HbA1c, for diabetes complications. In this study, we propose to investigate: (i) the time course of deterioration of physiological glucoregulatory mechanisms leading to increased GV, and (ii) the association of GV with metabolic and behavioral factors such as insulin sensitivity and treatment adequacy. Our primary hypothesis is:

Glucose variability in T1DM is triggered by behavioral events (e.g. meals, insulin injection, exercise) that challenge the metabolic system. The timing and the magnitude of the behavioral challenges, and the ability of the metabolic mechanisms to absorb these challenges, determine the magnitude of GV. This process develops in a certain time frame, and can be accelerated by inadequate treatment, or attenuated by precise timing and dosing of bio-behavioral control. This study will use a combination of treatment records, continuous glucose monitoring (CGM), and an inpatient admission to clarify the relationships between behavioral challenges to the metabolic system, physiological glucoregulatory mechanisms, and GV. This study will test the following hypotheses:

1. Suboptimal treatment behavior, e.g. insulin mistiming (early/late meal insulin) or unbalanced insulin (higher basal/bolus ratio), is correlated with higher GV and repeated hypo- and hyperglycemia; this relationship is mediated by a patients' insulin sensitivity;
2. A metabolic challenge (e.g. consecutive sequence of hypo- and hyperglycemia), will push the metabolic system into a transient super-critical state characterized by increased GV as defined by the Variability Grid Analysis (VGA) and the Average Daily Risk Range (ADRR), which will persist for several days beyond the discontinuation of the challenge.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes mellitus for ≥2 years. For an individual to be enrolled at least one criterion from each list must be met.

  * Criteria for documented hyperglycemia (at least 1 must be met):

    * Fasting Blood Glucose (BG) ≥126 mg/dL
    * 2h Oral Glucose Tolerance Test (OGTT) ≥200 mg/dL
    * Hemoglobin (HbA1c) ≥6.5%
    * BG ≥200 mg/dL with symptoms
    * History of hyperglycemia consistent with diabetes
  * Criteria for requiring insulin at diagnosis (1 must be met):

    * required insulin at diagnosis and continually thereafter
    * no insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and insulin eventually required and used continually
    * no insulin at diagnosis but continued hyperglycemia, positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and insulin eventually required and used continually
* Use of an insulin pump for at least six months prior to the study.
* Using a bolus calculator with pre-defined parameters for carbohydrate ratio(s), and insulin sensitivity factor(s).
* Signed informed consent.
* Age ≥21 and <65 years old.
* HbA1c ≤10% as measured with DCA 2000 or equivalent device.
* Willingness to use lispro (Humalog) insulin for metabolic challenge admission.
* Willingness to perform self-monitoring blood glucose (SMBG) >4 times/day.
* Willingness to avoid consumption of acetaminophen-containing products during the study.
* Willingness to perform 4 days of outpatient assessment with timed, prepackaged meals and snacks, and >7 SMBGs.

Exclusion Criteria:

* Uncontrolled arterial hypertension (resting blood pressure >160/100 mm Hg).
* Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥3 times the upper reference limit.
* Impaired renal function: glomerular filtration rate (calc GFR) of <60 ml/min/1.73 m2.
* Diabetic ketoacidosis in the past 6 months
* Conditions which may increase the risk of induced hypoglycemia such as:

  * uncontrolled coronary artery disease
  * stable or unstable angina
  * episode of chest pain of cardiac etiology with documented Electrocardiography changes or positive troponin levels
  * positive stress test
  * catheterization with coronary blockages >50%
  * congestive heart failure
  * significant cardiac arrhythmia
  * history of a cerebrovascular event
  * seizure disorder
  * syncope
  * adrenal insufficiency
  * hypoglycemia-induced migraine within the past year
  * neurological disease
* Diabetic complications altering insulin kinetics or food absorption
* Pregnancy, breast-feeding or intention of becoming pregnant.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment).
* skin condition that prevents sensor placement on the abdomen or arm.
* Difficulties to operate Continuous Glucose Monitor.
* Uncontrolled thyroid disease: thyroid-stimulating hormone (TSH)>10.
* Bleeding diathesis or dyscrasia.
* Alcohol or drug abuse within 1 year of enrollment by patient history.
* Allergy to components of the CGM sensor.
* Blood donation >473 ml in last 56 days
* Prior noncompliance with study procedures.
* Hematocrit outside of the normal range.
* Magnesium <1.6 mg/dl.
* Potassium <3.4 mmol/L.
* Active enrollment in another clinical trial
* Allergy to or intolerance of insulin lispro (Humalog)
* Anticoagulant therapy other than aspirin.
* Oral steroids.
* Use of acetaminophen-containing medication that cannot be.
* Use of Type 2 Diabetes Mellitus medications: including metformin, sulfonylureas, meglitinides, thiazolidinediones, Dipeptidyl peptidase-4 (DPP-IV) inhibitors, glucagonlike Peptide (GLP-1) agonists and alpha-glucosidase inhibitors.
* Unwillingness to withhold Pramlintide for the duration of the study intervention.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Breton, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from the Center's recruitment database.
Pre-assignment Details: Subject will be trained & wear a blinded CGM for 2 days. Data will be collected about diabetes management including blood glucose data from SMBG & CGM values along with insulin pump records throughout the 4 wk observation period. Subjects will then be admitted to the study unit for a metabolic challenge.
Groups:
- Glucose Variability Observation: The study procedures will start after CGM device training & practice using the blinded CGM for 2 days and will continue over the course of ~33 days. The study team will collect data about diabetes management including blood glucose data from fingerstick and CGM values along with insulin pump records throughout the 4 wk observation period. Insulin sensitivity will be evaluated at home with predetermined meals' carbohydrate count. At the mid-study point glucose variability (GV) will be simulated in clinic with a metabolic challenge (liquid mixed meal) followed 4h later by the induction of hypoglycemia with an intravenous insulin injection. Insulin sensitivity, as well as glucagon and epinephrine counterregulatory responses will be evaluated to be related to overall Glucose Variability.
  GV Observation: On the morning of ~Day 17 for a metabolic challenge involving a standardized liquid mixed meal intended to raise the blood glucose approximately 150 mg/dl, followed four hours la
Period: Overall Study
Arm/Group | Glucose Variability Observation
Started | 30
Training | 30
Observation Period | 28
Physiological Test | 28
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Glucose Variability Observation: The study procedures will start after CGM device training & practice using the blinded CGM for 2 days and will continue over the course of ~33 days. The study team will collect data about diabetes management including blood glucose data from fingerstick and CGM values along with insulin pump records throughout the 4 week observation period. Insulin sensitivity will be evaluated at home with predetermined meals' carbohydrate count. At the mid-study point glucose variability will be simulated in clinic with a metabolic challenge (liquid mixed meal) followed 4 hours later by the induction of hypoglycemia with an intravenous insulin injection. Insulin sensitivity, as well as glucagon and epinephrine counterregulatory responses will be evaluated to be related to overall Glucose Variability.
  Glucose Variability Observation: On the morning of ~Day 17 for a metabolic challenge involving a standardized liquid mixed meal, followed four hours later by the induction of hypoglycemia.
Arm/Group | Glucose Variability Observation
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change Between Pre and Post Challenge Glucose Variability
Description: Glucose variability in the days leading to and following the challenge was assessed by computing Low Blood Glucose Index (LBGI) on daily self-monitoring of BG (SMBG) readings. Low LBGI values correspond to lower glucose variability associated with hypoglycemic risk. LBGI values lie between 0 and 100
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Low Hypoglycemia Exposure (Group 1); Medium Hypoglycemia Exposure - Group 2; High Hypoglycemia Exposure - Group 3: To test the impact of prior exposure to low BG on the challenge effect on short-term glucose variability, the study participants were stratified in 3 different groups, based on the number of hypoglycemic episodes below 70 mg/dl they had experienced in the 2 weeks preceding the intervention. The groups were identified as follows: Group 1 - subjects who had experienced hypoglycemia once every 3 days or less, in the 2 weeks before the challenge (0 to 4 events); Group 2 - subjects who had experienced hypoglycemia approximately once every 2 days (5 to 9 events); Group 3 - subjects reporting approximately 1 or more hypoglycemic events per day (10 events or more).
Arm/Group | Low Hypoglycemia Exposure (Group 1) | Medium Hypoglycemia Exposure - Group 2 | High Hypoglycemia Exposure - Group 3
Number analyzed (Participants) | 10 | 8 | 10
score on a scale
  pre challenge | 0.51 [0.4 to 0.82] | 1.62 [1.01 to 2.14] | 3.71 [1.9 to 4.34]
  post challenge | 0.97 [0.46 to 1.39] | 1.9 [1.38 to 2.52] | 5.42 [3.41 to 6.51]

ADVERSE EVENTS:
Arm/Group | Glucose Variability Observation
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucose Variability Observation (N=30)
Sinus Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes